CLINICAL TRIAL: NCT00599781
Title: Treatment of ADA-SCID by Gene Therapy on Somatic Cells
Brief Title: Gene Therapy for ADA-SCID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Fondazione Telethon (Other)
Responsible Party: Claudio Bordignon, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150291
Record Dates: First submitted 2008-01-08; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2007-12

CONDITIONS: Severe Combined Immunodeficiency Syndrome
Keywords: adenosine deaminase; SCID; gene therapy; retroviral vector
MeSH Terms: conditions — Severe Combined Immunodeficiency | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PBL/HSC (Experimental)
  Interventions: Genetic: gene transduced PBL and/or gene transduced HSC

INTERVENTIONS:
Genetic: gene transduced PBL and/or gene transduced HSC — infusions of autologous PBL and/or HSC transduced with retroviral vectors encoding ADA
  Other Names: gene therapy

SUMMARY:
This study investigated the safety and efficacy of different gene therapy approaches for Severe Combined Immunodeficiency (SCID) caused by the deficiency of adenosine deaminase (ADA) enzyme. This is a severe condition that can be cured by HLA-matched sibling donor bone marrow transplantation. Patients were enrolled if no HLA-identical sibling donor was available and the patient showed evidence of failure of enzyme replacement therapy or this treatment was not a long-term available option. The aim of the study was to evaluate the safety and efficacy of the procedure and to identify the relative role of peripheral blood lymphocytes and hematopoietic stem cells and progenitor cells in the long-term reconstitution of immune functions after retroviral vector mediated ADA gene transfer.

DETAILED DESCRIPTION:
This is mono-centric, non-randomized, non-controlled, open label, phase I-II trial that evaluated the safety and efficacy of ADA gene transfer into somatic cells for the treatment of ADA-SCID

ELIGIBILITY:
Inclusion Criteria:

* Lack of HLA-identical sibling donor and
* Evidence of failure of the enzyme replacement treatment after >6 months or
* PEG-ADA is not available as a life long option

Exclusion Criteria:

* HLA identical bone marrow sibling donor
* HIV infection
* Malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1992-03; Primary Completion 2006-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety of the administration of the autologous PBL and/or autologous HSC transduced with the normal human ADA gene

SECONDARY OUTCOMES:
Evaluation of extent, kinetic and duration of the engraftment of transduced cells and the potential selective advantage of ADA positive cells
Evaluation of efficacy of the administration of autologous PBL/HSC(Clinical, immunological, hematological, microbiological, ADA activity and purine metabolism)
To identify the relative role of peripheral blood lymphocytes and hematopoietic stem cells and progenitor cells in the long-term reconstitution of immune functions after gene therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bordignon Claudio, MD, Principal Investigator — IRCCS San Raffaele

REFERENCES:
- [Derived] Sauer AV, Brigida I, Carriglio N, Hernandez RJ, Scaramuzza S, Clavenna D, Sanvito F, Poliani PL, Gagliani N, Carlucci F, Tabucchi A, Roncarolo MG, Traggiai E, Villa A, Aiuti A. Alterations in the adenosine metabolism and CD39/CD73 adenosinergic machinery cause loss of Treg cell function and autoimmunity in ADA-deficient SCID. Blood. 2012 Feb 9;119(6):1428-39. doi: 10.1182/blood-2011-07-366781. Epub 2011 Dec 19. PMID 22184407
- [Derived] Cassani B, Montini E, Maruggi G, Ambrosi A, Mirolo M, Selleri S, Biral E, Frugnoli I, Hernandez-Trujillo V, Di Serio C, Roncarolo MG, Naldini L, Mavilio F, Aiuti A. Integration of retroviral vectors induces minor changes in the transcriptional activity of T cells from ADA-SCID patients treated with gene therapy. Blood. 2009 Oct 22;114(17):3546-56. doi: 10.1182/blood-2009-02-202085. Epub 2009 Aug 3. PMID 19652199
- [Derived] Sauer AV, Mrak E, Hernandez RJ, Zacchi E, Cavani F, Casiraghi M, Grunebaum E, Roifman CM, Cervi MC, Ambrosi A, Carlucci F, Roncarolo MG, Villa A, Rubinacci A, Aiuti A. ADA-deficient SCID is associated with a specific microenvironment and bone phenotype characterized by RANKL/OPG imbalance and osteoblast insufficiency. Blood. 2009 Oct 8;114(15):3216-26. doi: 10.1182/blood-2009-03-209221. Epub 2009 Jul 24. PMID 19633200
- [Derived] Aiuti A, Cattaneo F, Galimberti S, Benninghoff U, Cassani B, Callegaro L, Scaramuzza S, Andolfi G, Mirolo M, Brigida I, Tabucchi A, Carlucci F, Eibl M, Aker M, Slavin S, Al-Mousa H, Al Ghonaium A, Ferster A, Duppenthaler A, Notarangelo L, Wintergerst U, Buckley RH, Bregni M, Marktel S, Valsecchi MG, Rossi P, Ciceri F, Miniero R, Bordignon C, Roncarolo MG. Gene therapy for immunodeficiency due to adenosine deaminase deficiency. N Engl J Med. 2009 Jan 29;360(5):447-58. doi: 10.1056/NEJMoa0805817. PMID 19179314
- [Derived] Cassani B, Mirolo M, Cattaneo F, Benninghoff U, Hershfield M, Carlucci F, Tabucchi A, Bordignon C, Roncarolo MG, Aiuti A. Altered intracellular and extracellular signaling leads to impaired T-cell functions in ADA-SCID patients. Blood. 2008 Apr 15;111(8):4209-19. doi: 10.1182/blood-2007-05-092429. Epub 2008 Jan 24. PMID 18218852